CLINICAL TRIAL: NCT03563742
Title: Open-Label Study With Rilpivirine in Treatment-naïve Indian Subjects With HIV-1 Infection to Determine Safety and Efficacy
Brief Title: A Study to Determine the Safety and Efficacy of Rilpivirine in Treatment-naive Indian Participants With Human Immunodeficiency Virus Type 1 (HIV-1) Infection
Acronym: RISE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: High SF rate (less treatment-naïve subjects & subjects with viral load <100000). Reevaluation in scientific position in India after internal discussion.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108402; TMC278HTX3001 (Other: Johnson & Johnson Pte Ltd)
Record Dates: First submitted 2018-05-28; First posted 2018-06-20 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Human Immunodeficiency Virus Infections
Keywords: Treatment-naive; rilpivirine; India
MeSH Terms: interventions — Rilpivirine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment: Rilpivirine+Combination Therapy (TDF/3TC) (Experimental): The participants will receive antiretroviral treatment of rilpivirine 25 milligram (mg) tablet orally once daily from Day 1 for 48 weeks with a meal to improve absorption. The participants will also receive background combination therapy of 1 tablet orally once daily containing 300 mg tenofovir disoproxil fumarate (TDF) and 300 mg lamivudine (3TC).
  Interventions: Drug: Rilpivirine 25 mg; Drug: Tenofovir Disoproxil Fumarate (TDF)/Lamivudine (3TC)

INTERVENTIONS:
Drug: Rilpivirine 25 mg — Participants will receive rilpivirine 25 mg tablet orally once daily.
  Other Names: Edurant
Drug: Tenofovir Disoproxil Fumarate (TDF)/Lamivudine (3TC) — Participants will receive 1 fixed dose combination tablet once daily containing 300 mg TDF and 300 mg 3TC.
  Other Names: Tenvir-L

SUMMARY:
The primary purpose of the study is to evaluate the efficacy of rilpivirine (RPV)-based regimen in human immunodeficiency virus type 1 (HIV-1) infected, antiretroviral (ARV) treatment-naive participants, as determined by the percentage of virologic responders defined as having HIV-1 ribonucleic acid (RNA) less than 400 copies/ milliliter (mL) at Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Must have documented human immunodeficiency virus type 1 (HIV-1) infection
* Must be antiretroviral (ARV) treatment-naïve
* Have plasma HIV-1 ribonucleic acid (RNA) less than (<) 100,000 copies/milliliter (mL) at screening visit
* Have cluster of CD4+ T-cell count (greater than) >200/ cubic millimeter (mm^3) at screening visit
* Women of childbearing potential must have a negative serum (beta human chorionic gonadotropin [beta hCG]) pregnancy test at screening; and a negative urine (or serum, if required by local regulations) pregnancy test before the first dose of study

Exclusion Criteria:

* History of any primary nucleo(t)side reverse transcriptase inhibitor (N[t]RTI) or non-nucleoside reverse transcriptase inhibitor (NNRTI) mutations (if testing performed locally, and results are available), as defined by the current International AIDS (acquired immunodeficiency syndrome) Society-United States (USA) (International Antiviral Society-USA) 2017 guidelines
* Has clinical or laboratory evidence of significantly decreased hepatic function or decompensation, irrespective of liver enzyme levels (hepatic insufficiency)
* Diagnosed with acute viral hepatitis at screening or before baseline
* Infected with Mycobacterium tuberculosis which is likely to require rifampicin-based treatment during the study
* Has a Grade 3 or 4 laboratory abnormality as defined by the Division of AIDS (DAIDS) for Grading the Severity of Adult and Pediatric Adverse Events criteria with the following exceptions unless clinical assessment foresees an immediate health risk to the participant: (a) Preexisting diabetes or with asymptomatic glucose Grade 3 or 4 elevations (b) Asymptomatic triglyceride or cholesterol elevations of Grade 3 or 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who are Virologic Responders (HIV-1 RNA <400 Copies/mL) at Week 24 | Week 24
  Virologic responders are defined as participants having viral load (plasma Human Immunodeficiency Virus-Type 1 Ribonucleic Acid [HIV-1 RNA] levels) less than (<) 400 copies/milliliter (mL) at Week 24 (Food and Drug Administration [FDA]-defined snapshot analysis).

SECONDARY OUTCOMES:
Percentage of Participants who are Virologic Responders (HIV-1 RNA <50 Copies/mL) at Week 24 | Week 24
  Virologic responders are defined as participants having viral load (plasma HIV-1 RNA levels) <50 copies/mL at Week 24 (FDA-defined snapshot analysis).
Percentage of Participants who are Virologic Responders (Plasma HIV-1 RNA Levels <50, <400 and <1,000 Copies/mL) at Week 48 | Week 48
  Virologic responders are defined as participants having viral load (plasma HIV-1 RNA levels) <50, <400 and <1,000 copies/mL at Week 48 (FDA-defined snapshot analysis).
Absolute Value in Cluster of Differentiation 4 Positive (CD4+) T-Cell Count at Weeks 24 and 48 | At Weeks 24 and 48
  CD4+T cell absolute counts will be determined at Weeks 24 and 48.
Change from Baseline in CD4+ T Cell Count at Weeks 24 and 48 | Baseline, Weeks 24 and 48
  Change from baseline in CD4+ T cell count will be determined at Weeks 24 and 48.
Percentage of Participants with Grade 3 and 4 Adverse Events (AEs), Serious Adverse Events (SAEs), and Participants Experiencing Premature Discontinuation due to AEs Through Week 48 | Through Week 48
  Percentage of participants with Grade 3 and 4 AEs will be assessed. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Percentage of participants who prematurely discontinued study due to AEs will also be analyzed.
Percentage of Participants with Laboratory Abnormalities | Up to Week 48
  Percentage of participants with laboratory abnormalities will be reported.
Number of Participant with Clinically Significant Change from Baseline in Laboratory Parameters | Baseline up to Week 48
  Number of participants with clinically significant change from baseline in laboratory parameters related to hematology, serum chemistry will be assessed.
Emergence of Viral Resistance Through Weeks 24 and 48 | Through Weeks 24 and 48
  Resistance analysis will be determined using genotypic analysis at the time of virological failure (that is, 2 consecutive plasma HIV-1 RNA levels greater than or equal to [>=] 400 copies/mL through Weeks 24 and 48 of study treatment).
Percentage of Participant with Treatment Adherence (95%) Based on Tablet Count up to Weeks 24 and 48 | Up to Weeks 24 and 48
  Percentage of adherent participants as measure of treatment compliance will be assessed by tablet count.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- India (5):
  - Chennai Antiviral Research and Treatment(CART) Clinical Research Site, Chennai
  - YRGCARE, Chennai
  - Manipal University-Kasturba Medical College, Mangalore
  - Lata Mangeshkar Hospital, Nagpur
  - Deenanath Mangeshkar Hospital and Research Centre, Pune

REFERENCES:
- See also: Open-Label Study with Rilpivirine in Treatment-naïve Indian Subjects With HIV-1 Infection to Determine Safety and Efficacy — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108402&attachmentIdentifier=a3a0582b-a3a9-45e7-91c8-b42f2cbb4e6d&fileName=CR108402_CSR_Synopsis.pdf&versionIdentifier=